CLINICAL TRIAL: NCT02108444
Title: Hepatitis B Virus Reactivation After Withdrawal of Prophylactic Antiviral Therapy in Lymphoma Patients With Hepatitis B Virus Infection
Brief Title: Hepatitis B Virus Reactivation After Withdrawal of Prophylactic Antiviral Therapy in Lymphoma Patients
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Chairman of lymphoma department, Peking University
Other Study IDs: PKU 2013-Autonomous-9
Record Dates: First submitted 2014-03-30; First posted 2014-04-09 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Hepatitis; Hepatitis B; Lymphoma; Hematologic Diseases
Keywords: hepatitis; hepatitis B; lymphoma; Hematologic Diseases
MeSH Terms: conditions — Hepatitis; Hepatitis B; Lymphoma; Hematologic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — serum hepatitis B virus DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group with HBV reactivation: group with hepatitis B virus reactivation
- group without HBV reactivation: group without hepatitis B virus reactivation

SUMMARY:
This study is a retrospective analysis to explore the incidence of hepatitis B virus reactivation after withdrawal of prophylactic antiviral therapy, the efficacy and safety of chemotherapy, and overall survival rate in lymphoma patients with hepatitis B virus infection.

DETAILED DESCRIPTION:
All eligible patients received prophylactic antiviral therapy during and within 6 months after chemotherapy in previous sudy. We did not assign specific interventions to the subjects in this study. The primary endpoint of this study is the incidence of hepatitis B virus reactivation after withdrawal of prophylactic antiviral therapy. The secondary endpoints include the incidence of hepatitis flare related to hepatitis B virus reactivation after withdrawal of prophylactic antiviral therapy, the tumor response rate, and overall survival rate.

ELIGIBILITY:
Inclusion Criteria:

* treatment-naive patients with lymphoma
* patients with a history of previous exposure to hepatitis B virus (HBV): HBsAg or hepatitis B core antibody (anti-HBc) positive

Exclusion Criteria:

* HBsAg and HBcAb negative

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lymphoma patients with hepatitis B virus infection diagnosed in Peking University Cancer Hospita
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2007-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
the incidence of hepatitis B virus delayed reactivation | within one year after withdrawal of prophylactic antiviral therapy
  hepatitis B virus reactivation after withdrawal of prophylactic antiviral therapy

SECONDARY OUTCOMES:
the incidence of hepatitis B virus related hepatitis flare | within one year after withdrawal of prophylactic antiviral therapy
  the incidence of hepatitis B virus related hepatitis flare after withdrawal of prophylactic antiviral therapy
Number of patients that achieve a tumor response | within one year after withdrawal of prophylactic antiviral therapy
overall survival rate | within one year after withdrawal of prophylactic antiviral therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD., Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China